CLINICAL TRIAL: NCT06354868
Title: A Prospective Observational Clinical Study to Investigate the Relationship Between Seizure Frequency and BioEP During ASM Titration in Newly Diagnosed Patients With Epilepsy, and to Assess the Utility of BioEP as an Early Prognostic Indicator of Anti-seizure Medication (ASM) Efficacy
Brief Title: A Study to Assess utiLity of BIoEP as an Early Prognostic Indicator for Predicting Anti-Seizure Medication (ASM) Efficacy
Acronym: ECLIPSE
Status: Not yet recruiting | Type: Observational
Sponsor: Neuronostics Ltd (Industry)
Collaborators: Cornwall Partnership NHS Foundation Trust (Network)
Responsible Party: Sponsor
Other Study IDs: NNBioEP004
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multisite prospective clinical study is to investigate the relationship between seizure type and frequency with the BioEP result during ASM titration in newly diagnosed patients with epilepsy, and to assess the utility of BioEP as an early prognostic indicator of ASM efficacy

DETAILED DESCRIPTION:
The study will consist of a cohort of adult patients who present to first seizure clinics. The patients will have had an EEG performed as part of the clinical care pathway (this will act as their baseline reference BioEP value). They will also have received an epilepsy diagnosis and will be due to start ASM titration as part of their epilepsy treatment. One stop clinics shall be targeted primarily for their same day EEGs service, to allow a baseline EEG to be obtained prior to the patient starting ASMs in those who get an EEG diagnosis on the same day.

Patients who have initially seen a Neurologist in a first seizure clinic and are under a period of watchful waiting, and then return to the clinic a second time and receive an epilepsy diagnosis will be eligible to enter the trial. The second encounter with Neurology would usually be due to the occurrence of a second seizure or by a positive EEG being recorded as part of their usual care during the watch and wait period and the clinician deciding to start ASMS on that basis. The study will utilise their 1st EEG performed as the baseline EEG (provided this is performed within a 12-month window prior to their second Neurology encounter and during a period of no ASMs).

A baseline BioEP result shall be gathered from baseline EEG data prior to commencement of the ASM titration regime and a set of computational biomarkers (BioEP) shall be identified from relevant EEG segments free of IEDs. In addition to the clinical care pathway, participants will also receive additional routine EEGs at 1, 3 and 6 and 12 months after commencing treatment. The EEGs performed at 1, 3, 6 and 12 months duration shall also have their BioEP results identified at these specified time points.

Any patient who requires a ASM medication change during the first 6 months of the trial, an additional EEG will be collected at 9 months, and then again at the usual 12 months' time point.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and above) presenting with first suspected seizure(s).
* Able to give informed consent.
* Patient has received an initial epilepsy diagnosis.
* Patient accepts decision to commence ASM.
* Have an EEG prior to commencing ASMs.
* Participants under watchful waiting who subsequently return to clinic for an epilepsy diagnosis (following a second seizure or a positive EEG) can be included in the study. They must have had an EEG performed in the 12 months prior to be being included in the study (to be used as a baseline EEG) and not have been taking any ASMs at the time.

Exclusion Criteria:

* Participants unable to tolerate an EEG test so no EEG data were gathered.
* Participants with a known hepatic/renal encephalopathy.
* Patient diagnosed with possible NEAD and epilepsy (dual diagnosis).
* Participants taking part in another Clinical Trial of an Investigational Medicinal Product (CTIMP) (qualitative/observational studies are acceptable).
* Patient receiving low does ASMs for other conditions (migraines etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the first seizure clinic, receive a routine EEG, receive a diagnosis of epilepsy and are commenced an ASM.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The relationship between BioEP and seizure frequency. | 12 months
  Identify a ratio of change of BioEP result from baseline (prior to ASMs commencing) to maximal effects of the ASM intervention and seizure control.

SECONDARY OUTCOMES:
Association between the 12-month change from baseline in BioEP result and the patients reported global impression of change | 12 months
  The investigators will examine the association between the 12-month change from baseline in BioEP score and reporting at least 'a little improved' on the 7-point patient global impression of change scale. Minimum value 1 = very much improved, maximum value 7 = very much worse A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Milaana Mainstone, Study Director — Neuronostics Ltd